CLINICAL TRIAL: NCT02391441
Title: Imaging of Ventricular Reversed Remodeling After Double Lung Transplantation in Patients With Pulmonary Arterial Hypertension
Brief Title: Ventricular Reversed Remodeling After LTX in PAH Patients
Acronym: PAH-LTX
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, J.P. van Melle, MD PhD, University Medical Center Groningen
Other Study IDs: METc2014/134
Record Dates: First submitted 2015-03-06; First posted 2015-03-18 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary; Arterial; Hypertension; Lung; Transplantation; MRI
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pulmonary arterial hypertension: Patients who are on the waiting list for double-LTX for pulmonary arterial hypertension.
- Control group: Control patients without increased pulmonary artery pressure (i.e. RV peak pressure <35 mmHg measured with echocardiography) who are on the waiting list for double-LTX.

SUMMARY:
The investigators will evaluate ventricular reversed remodelling after double lung transplantation (LTX) in patients with pulmonary arterial hypertension (PAH), measured with cardiac magnetic resonance imaging (MRI). Reversed remodelling will be compared with control patients without PAH (e.g. Cystic Fibrosis) who will also undergo LTX.

DETAILED DESCRIPTION:
In this study, pre-LTX and six-months post-LTX measurements will be compared with each other and between the primary and control group.

Pre- and post-LTX measurements include:

Past medical history: Including basic diagnosis; interventions, surgery and transplant related complications (re-operations, hospitalizations, infections) and medication history; These data will be collected by studying the medical files including surgical reports.

Present medical history: Including NYHA class.

Physical examination: Including length and weight.

Cardiac Magnetic Resonance Imaging:

* Ventricular volume, function and mass measurements
* Flow measurements of the pulmonary artery and aorta
* Disease specific measurements (e.g. septal bowing, RV trabecularisation, etc.)
* T1-mapping

Transthoracic Echocardiography

Resting ECG: Disease specific electrophysiological findings (e.g. QRS-duration, right bundle branch block).

Laboratory evaluation:

* NT-pro-BNP
* eGFR
* Remaining serum will be stored.

ELIGIBILITY:
Inclusion criteria:

* Patients who are on the waiting list for double-LTX, in our institution, for pulmonary arterial hypertension.
* Eligible for CMR imaging
* No claustrophobia
* No pacemaker, ICD, etc.
* Informed consent

Exclusion criteria:

* Inability to comply with primary endpoint measures.
* Body mass index ≥40 kg/m2.
* Pregnant patients will not be included, they may be included >3 months after pregnancy.
* Patients with age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary arterial hypertension and control patients without increased pulmonary artery pressure who are on the waiting list for double-LTX
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-03; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Ventricular remodeling on cardiac magnetic resonance | Six months postoperative
  Absolute increase in RV ejection fraction
Ventricular remodeling on cardiac magnetic resonance | Six months postoperative
  Absolute increase in LV ejection fraction
Ventricular remodeling on cardiac magnetic resonance | Six months postoperative
  Absolute decrease in RV myocardial mass
Ventricular remodeling on cardiac magnetic resonance | Six months postoperative
  Absolute increase in LV myocardial mass
Ventricular remodeling on cardiac magnetic resonance | Six months postoperative
  Absolute decrease in RV end-diastolic volume
Ventricular remodeling on cardiac magnetic resonance | Six months postoperative
  Absolute increase in LV end-diastolic volume
Ventricular remodeling on cardiac magnetic resonance | Six months postoperative
  Restoration of septal displacement
Ventricular remodeling on cardiac magnetic resonance | Six months postoperative
  Decrease in RV myocardial extracellulair volume assessed with T1-mapping
Ventricular remodeling on cardiac magnetic resonance | Six months postoperative
  Decrease in LV end-systolic eccentricity index

SECONDARY OUTCOMES:
Functional remodeling patterns after LTX, assessed with echocardiography | Six months postoperative
  Increase in tricuspid annular plane systolic excursion (i.e. TAPSE)
Functional remodeling patterns after LTX, assessed with echocardiography | Six months postoperative
  Increase in myocardial performance index (MPI) or Tei index
Functional remodeling patterns after LTX, assessed with echocardiography | Six months postoperative
  Increase in tricuspid annular systolic motion velocity (i.e. RV s')
Functional remodeling patterns after LTX, assessed with echocardiography | Six months postoperative
  Increase in RV (global/septal/free wall) longitudinal strain
Functional remodeling patterns after LTX, assessed with echocardiography | Six months postoperative
  Decrease in RA size
Functional remodeling patterns after LTX, assessed with echocardiography | Six months postoperative
  Increase in LA size
Change in heart failure biomarkers | Six months postoperative
  Decrease in NT pro-BNP
Electrocardiographic remodeling | Six months postoeprative
  Normalization of RV hypertrophy and strain
Electrocardiographic remodeling | Six months postoeprative
  Normalization of right axis deviation
Electrocardiographic remodeling | Six months postoeprative
  Normalization of right atrial enlargement

OTHER OUTCOMES:
Functional outcome | Six months postoperative
  Decrease in NYHA-class

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J van Veldhuisen, MD PhD, Study Director — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands